CLINICAL TRIAL: NCT04490369
Title: Evaluation of Pain and Discomfort in the Cardiac Catheterization Lab
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102686
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-01

CONDITIONS: Patient Comfort
Keywords: Procedural sedation; Cardiac Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1- short interval: Less than or equal to six minutes between receiving sedation and the start of the procedure
- Group 2- long interval: Greater than or equal to seven minutes between receiving sedation and the start of the procedure

SUMMARY:
The purpose of this study is to explore how the timing of procedural sedation medications influences patient comfort and satisfaction with sedation.

Participation in this study will included be randomly assigned to one of two groups (long and short) within standard of care. Each group will observe a time interval between receiving procedural sedation medications and the start of the procedure. A trained observer will evaluate patient experience during the procedure and at the end of the procedure we will ask the participant 3 brief questions about the experience. All other information collected about the experience during the procedure will occur as part of usual care. No further activities will be asked as part of this study. All study activities will occur during a scheduled visit and participation is complete once questions have been answered.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Coming to Duke University for Cardiac Catheterization

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients coming to Duke University for Cardiac Catheterization
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Total medication administration dosage as measured by the procedural database | During procedure, up to 2.5 hours
Frequency of medication administration as measured by the procedural database | During procedure, up to 2.5 hours

SECONDARY OUTCOMES:
Patient satisfaction as measured by Procedural Sedation Assessment Survey (PROSAS) | Within 2 hours of procedure
Pain as measured by observation using the Behavioral Pain Assessment Tool (BPAT) | During procedure, to 2.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bradi Granger, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mall A, Girton TA, Yardley K, Ronn M, Cross E, Smith PJ, Rossman P, McEwen T, Ohman EM, Jones WS, Granger BB. Timing of sedation and patient-reported pain outcomes during cardiac catheterization: Results from the UNTAP-intervention study. Catheter Cardiovasc Interv. 2023 Jan 14. doi: 10.1002/ccd.30535. Online ahead of print. PMID 36640418